CLINICAL TRIAL: NCT02009709
Title: Study of the Safety and Effectiveness of Photochemically Induced Collagen Cross-Linking at an Irradiance of 9 mW/cm2 and 18 mW/cm2 in Eyes With Keratoconus or Ectasia
Brief Title: Study of the Safety and Effectiveness of Collagen Cross-Linking at an Irradiance of 9 mW/cm2 and 18 mW/cm2
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Robert Mack, M.D. (Other)
Responsible Party: Sponsor-Investigator, Robert Mack, M.D., Sponsor-Investigator, Mack Eye Center
Organization: Mack Eye Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC-0001
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Keratoconus; Corneal Ectasia
Keywords: keratoconus; collagen crosslinking; crosslinking; ectasia
MeSH Terms: conditions — Keratoconus; Dilatation, Pathologic | interventions — Riboflavin; Ophthalmic Solutions; Chromatin Immunoprecipitation Sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 9 mW/cm2 (Active Comparator): CCL-VARIO UV lamp Riboflavin 0.1% ophthalmic solution
  Interventions: Drug: Riboflavin 0.1% ophthalmic solution; Device: CCL-VARIO UV lamp
- 18 mW/cm2 (Active Comparator): CCL-VARIO at 18 mW/cm2 Riboflavin 0.1% ophthalmic solution
  Interventions: Drug: Riboflavin 0.1% ophthalmic solution; Device: CCL-VARIO at 18 mW/cm2

INTERVENTIONS:
Drug: Riboflavin 0.1% ophthalmic solution — Instillation of 0.1% riboflavin ophthalmic solution, one drop every 3 minutes for 30 minutes before the procedure and one drop every 3 minutes during the procedure.
  Other Names: CXL; CCL; crosslinking
Device: CCL-VARIO UV lamp — Application of ultraviolet light on the eye to be treated at an irradiance of 9 mW/cm2 for 10 minutes
  Other Names: CXL; CCL; crosslinking
  Arms: 9 mW/cm2
Device: CCL-VARIO at 18 mW/cm2 — Application of ultraviolet light on the eye to be treated at an irradiance of 18 mW/cm2 for 5 minutes.
  Other Names: CXL; CCL; crosslinking
  Arms: 18 mW/cm2

SUMMARY:
The primary objective of this study is to determine the effectiveness and safety of corneal collagen cross-linking at irradiance levels of 9 and 18 mW/cm2.

ELIGIBILITY:
General Inclusion Criteria

Prospective subjects must meet all of the following criteria to be eligible for participation:

* 18 years of age or older
* Signed written informed consent
* Willingness and ability to comply with schedule for follow-up visits
* Contact lens removal prior to evaluation and treatment

Inclusion criteria for progressive keratoconus

Prospective subjects must meet two of the following criteria:

* Having a diagnosis of progressive keratoconus:
* An increase of ≥ 1.00 D in the steepest keratometry value
* An increase of ≥ 1.00 D in astigmatism manifest refraction
* A myopic shift (decrease in the spherical equivalent) of ≥ 0.50 D on subjective manifest refraction
* Presence of central or inferior steepening on the Pentacam map.
* Axial topography consistent with keratoconus
* Steepest keratometry (Kmax) value ≥ 47.00 D

Inclusion criteria for ectasia

Prospective subjects must meet the following criteria:

* History of having undergone a keratorefractive procedure
* Meeting two of the following criteria
* Steepening by topography, either Pentacam or Humphrey
* Thinning of cornea
* Shift in the position of thinnest portion of cornea
* Change in refraction with increasing myopia
* Development of myopic astigmatism
* Development of irregular astigmatism
* Loss of best spectacle corrected acuity. 6.2 Exclusion Criteria

Subjects meeting any of the following criteria will be excluded from this protocol:

* Eyes classified as either normal, atypical normal,
* Corneal pachymetry ≤ 350 microns at the thinnest point measured by Pentacam in the eye to be treated
* A history of chemical injury or delayed epithelial healing in the eye to be treated.
* Pregnancy (including plan to become pregnant) or lactation during the course of the study
* A known sensitivity to study medications
* Patients with nystagmus or any other condition that would prevent a steady gaze during the treatment
* Inability to cooperate with diagnostic tests.
* Patients with a current condition that, in the investigator's opinion, would interfere with or prolong epithelial healing.
* Taking Vitamin C (ascorbic acid) supplements within 1 week of the cross-linking treatment.
* Patients who are unable to remain supine and tolerate a lid speculum for an extended period of time.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Decrease in maximum corneal curvature | 3 and 6 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Mack, M.D., Principal Investigator — Mack Eye Center
Locations (1):
- Mack Eye Center, Hoffman Estates, Illinois, United States